CLINICAL TRIAL: NCT03119376
Title: Evaluation of an Online Tool (COBPeer) Dedicated to Junior Peer Reviewers for Assessing the Reporting of Randomized Controlled Trial Reports
Brief Title: Web-based Tool to Improve the Assessment of Reporting (COBPeer)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Oxford (Other); University of Ottawa (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Isabelle BOUTRON, Professor, Assistance Publique - Hôpitaux de Paris
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AC001
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Peer Review
Keywords: peer review; online tool; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- USUAL PEER REVIEWER (No Intervention): Two researchers will read all the peer-review reports and editors' comments for the first round. The researchers will determine whether the peer-reviewers and/or editors raised some concern on the completeness of reporting of the 10 CONSORT items considered and identified a switch primary outcome(s) between the manuscript and the register. The assessment of all peer-review reports and editors' comments for each manuscript will be combined (i.e., the item will be rated as incompletely reported if at least one peer reviewer rated it as such). The 2 researchers will be blinded to the gold standard assessment.
- COBPeer (Experimental): Junior peer reviewers will be invited to participate in an online training course on peer review (COBPeer).
  Interventions: Other: COBPEER
- GOLD STANDARD (No Intervention): Pairs of systematic reviewers will independently extract data from eligible reports. Reviewers involved in the data extraction will have expertise in the conduct of systematic reviews and will assess the completeness of reporting from the systematic reviewer perspective. They will not have access to the tool to avoid being influenced by the tool. The systematic reviewers will also systematically compare the primary outcome(s) reported in the manuscript and the primary outcome(s) reported in the registry and will document any discrepancies.

INTERVENTIONS:
Other: COBPEER — At the end of the online training, they can participate in the study and so peer review 1 manuscript randomly selected from our sample with our tool (COBPeer).
  Arms: COBPeer

SUMMARY:
The peer review process is a cornerstone of biomedical research publication. Despite being essential, the assessment of the completeness of the reporting and the identification of switched outcomes are not appropriately performed. Furthermore, these tasks do not suppose a high level of expertise and could be performed by junior researchers.

To assess the completeness of reporting and identified switched outcome(s), junior peer reviewers could use a simple online tool (COBPeer) based on the CONSORT (Consolidated Standards of Reporting Trials) 2010 checklist and Elaboration and Explanation publication for reporting parallel-group RCTs. The tool would feature bullet points eliciting the meaning of each checklist item. The aim of this study that will compare the accuracy of junior peer reviewers using the tool to that of usual peer reviewers when evaluating the completeness of reporting and switched of primary outcome(s) in reports of RCTs

DETAILED DESCRIPTION:
BACKGROUND: Context Inadequate reporting is a frequent cause of waste of research. To overcome this issue, the CONSORT statement, an evidence-based, minimum set of recommendations for reporting RCTs was developed in 1996. These guidelines have since been updated in 2001 and more recently in 2010. Many journals endorse the CONSORT statement. Some journals provide recommendations to authors to follow the CONSORT guidelines and some editors enforce the use of the CONSORT guidelines by requesting authors to submit a checklist in either the submission or acceptance stage. Nevertheless, inadequate reporting remains.

HYPOTHESE: To assess the completeness of reporting, junior peer reviewers could use a simple online tool based on the CONSORT 2010 checklist and Elaboration and Explanation publication for reporting parallel-group RCT

OBJECTIVE: 1) Develop an online tool and training module dedicated to junior peer reviewers for a) assessing the completeness of reporting of key items and b) identifying switched primary outcome(s) in reports of RCTs. 2) Compare the performance of junior peer reviewers using this tool with the usual peer-review process in identifying inadequate reporting and switched primary outcome(s) in reports of RCTs.

STUDY DESIGN: randomized ratio 1:1 controlled trial with two parallel arms. Participants will be invited to participate by invitation.

ELIGIBILITY: eligible participants are juniors peer reviewers. Junior peer reviewers are defined as early stage researchers: master students, PhD students, residents involved in clinical research during their study, and clinicians who have never reviewed a manuscript

INTERVENTION: the peer-review tool will be based on 10 items of the CONSORT Statement. This tool reminds the peer reviewer of the CONSORT item which must be reported by explicating it with a series of questions. The training module will explain each item to be evaluated with examples followed by a series of exercises from published randomized trial extracts.

MANUSCRIPT SELECTION: sample of randomized controlled trials published by Annals of Emergency Medicine, British Medical Journal, British Medical Journal Open and BioMed Central series medical.

EVALUATION BY THE JUNIOR PEER REVIEWERS: the junior peer reviewer who has accepted to participate and who has passed the training with success, will have to evaluate 1 article of the selected randomized sample.

EVALUATION OF THE USUAL PEER REVIEWERS: the evaluation by the usual peer-reviewers will be obtained by an analysis of the comments of the peer-reviewers which are available on line or obtained from the publisher.

GOLD STANDARD: peers of researchers who are experts in conducting systematic reviews will evaluate each article independently from other evaluations. Disagreements will be resolved by consensus.

PRIMARY OUTCOME: the mean number of items accurately classified per manuscript

SECONDARY OUTCOMES: the mean number of items accurately classified per manuscript for the 10 CONSORT items; the sensitivity, specificity and likelihood ratio to detect the item as adequately reported and to identify switch in primary outcome(s).

SAMPLE SIZE: 120 manuscripts and 120 peer reviewers juniors.

ELIGIBILITY:
Inclusion Criteria:

* master students,
* PhD students,
* residents involved in clinical research during their study,
* clinicians who have never reviewed a manuscript

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
the mean number of items accurately classified per manuscript | through study completion, an average of 6 month
  Each item will be classified as"adequately reported" (yes/no)

SECONDARY OUTCOMES:
the mean number of items accurately classified per manuscript for the 10 CONSORT items | through study completion, an average of 6 month
  Each item will be classified as"adequately reported" (yes/no)
the sensitivity, specificity and likelihood ratio to detect the item as adequately reported and to identify switch in primary outcome(s). | through study completion, an average of 6 month
  test for pair proportion

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu, 1, place du parvis de notre dame, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chauvin A, Ravaud P, Moher D, Schriger D, Hopewell S, Shanahan D, Alam S, Baron G, Regnaux JP, Crequit P, Martinez V, Riveros C, Le Cleach L, Recchioni A, Altman DG, Boutron I. Accuracy in detecting inadequate research reporting by early career peer reviewers using an online CONSORT-based peer-review tool (COBPeer) versus the usual peer-review process: a cross-sectional diagnostic study. BMC Med. 2019 Nov 19;17(1):205. doi: 10.1186/s12916-019-1436-0. PMID 31744489
- [Derived] Chauvin A, Moher D, Altman D, Schriger DL, Alam S, Hopewell S, Shanahan DR, Recchioni A, Ravaud P, Boutron I. A protocol of a cross-sectional study evaluating an online tool for early career peer reviewers assessing reports of randomised controlled trials. BMJ Open. 2017 Sep 15;7(9):e017462. doi: 10.1136/bmjopen-2017-017462. PMID 28918414